CLINICAL TRIAL: NCT03528499
Title: Scapular Movement Training Versus General Exercises for Individuals With Shoulder Pain: Randomized Controlled Trial
Brief Title: Scapular Movement Training Versus General Exercises for Individuals With Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Responsible Party: Principal Investigator, Danilo Harudy Kamonseki, Ms, PT, Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 86974318.7.0000.5504
Record Dates: First submitted 2018-04-23; First posted 2018-05-17 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Shoulder Pain; Musculoskeletal Disease; Joint Disease; Shoulder Injury
Keywords: Scapula; Physical Therapy; Movement; Rehabilitation
MeSH Terms: conditions — Shoulder Pain; Musculoskeletal Diseases; Joint Diseases; Shoulder Injuries | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scapular Movement Training (Experimental): Orientation and scapular exercises, performed twice a week, for 8 weeks.
  Interventions: Other: Scapular Movement Training
- General Exercises (Active Comparator): Scapulothoracic muscle stretching and strengthening exercises, performed twice a week, for 8 weeks.
  Interventions: Other: General Exercises

INTERVENTIONS:
Other: Scapular Movement Training — Orientation about the proper scapular position and movement and training to modify the scapular movement pattern.
  Other Names: Orientation and training
  Arms: Scapular Movement Training
Other: General Exercises — Strengthening and stretching exercises.
  Other Names: Exercises
  Arms: General Exercises

SUMMARY:
Interventions focused on the scapula have been frequently used to treat shoulder pain. However, most studies do not assess the contribution of scapular movement alteration for the symptoms.

Objectives: To compare the effects of two interventions for shoulder pain: Scapular Movement Training and General Exercises.

DETAILED DESCRIPTION:
This is a double-blinded randomized controlled trial. Sixty-four subjects with shoulder pain, scapular dyskinesis, and positive scapular assistance test will be randomized in two groups: 1) Scapular Movement Training, and 2) General Exercises. The Scapular Movement Training Group will receive the orientation about proper scapular position and movement, and will be trained to modify the scapular movement pattern. The General Exercises Group will perform scapulothoracic stretching and strengthening exercises.

Both groups will be treated twice a week for eight weeks. The following outcomes will be collected at baseline and follow-up: scapular kinematics, electromyographic muscle activity of the upper, middle and lower trapezius, and serratus anterior, as well as pain intensity, function, and fear avoidance beliefs. Also, pain intensity, function, and fear-avoidance beliefs will be assessed at the fourth week of follow-up after the end of treatment's period.

ELIGIBILITY:
Inclusion Criteria:

* Shoulder pain intensity ≥ 3 points on Numerical Rating Scale;
* Shoulder pain lasting ≥ 3 months;
* Scapular dyskinesis;
* Positive Scapular Assistance Test;
* Arm elevation ≥ 150°;

Exclusion Criteria:

* Body Mass index > 28Kg/m
* History of humerus, clavicle and scapula fracture and/or surgery;
* History of rotator cuff surgery or tears, shoulder dislocation, and instability;
* Frozen Shoulder;
* Neurological or systemic disease which may alter the muscle strength and sensibility;
* Positive Upper Limb Tension Test and/or Spurling's test
* Pregnancy;
* Physical therapy within 6 months;
* Corticosteroid injection within 3 months
* Transpore tape allergy;

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2018-08-21 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Change in Three-Dimensional Scapular Kinematics from baseline to 8 weeks. | Pre (baseline) and post Treatment (8 weeks)
  3-D Scapular kinematics (upward/downward rotation; internal/external rotation; anterior/posterior tilt) will be measured by an electromagnetic tracking system (in degrees).

SECONDARY OUTCOMES:
Change in Muscle activity from baseline to 8 weeks. | Pre (baseline) and post Treatment (8 weeks)
  Surface electromyographic recorded from scapulothoracic muscles (Upper trapezius, Middle Trapezius, Lower Trapezius and Serratus Anterior).
Change in Pain from baseline to follow-up. | Pre (baseline), 4 weeks, post Treatment (8 weeks), and follow-up (4 weeks after treatment )
  The pain will be measured with 11 point - Numerical Rating Pain Scale with scores ranging from 0 (no pain) to 10 (maximum pain).
Change in Function from baseline to follow-up. | Pre (baseline), 4 weeks, post Treatment (8 weeks), and follow-up (4 weeks after treatment )
  The Function will be measured with Disabilities of the Arm, Shoulder and Hand with scores ranging from 0 to 100 (higher score reflects greater disability).
Change in Fear-Avoidance Beliefs from baseline to follow-up. | Pre (baseline), 4 weeks, post Treatment (8 weeks), and follow-up (4 weeks after treatment )
  The Fear-Avoidance Beliefs Questionnaire (FABQ) contains 2 scales: FABQ work scale (with range from 0 to 42) and FABQ physical activity scale (with range from 0 to 24). Higher scores indicate higher levels of fear-avoidance beliefs.
Change in Overall improvement of Symptoms from baseline to follow-up. | Pre (baseline), 4 weeks, post Treatment (8 weeks), and follow-up (4 weeks after treatment )
  The Overall improvement of Symptoms will be measured with the Global Rating of Change Scale with scores ranging from -7 to +7 (A higher score indicates higher recovery from the condition).
Change in Kinesiophobia from baseline to follow-up | Pre (baseline), 4 weeks, post Treatment (8 weeks), and follow-up (4 weeks after treatment )
  The Kinesiophobia will be measured with Tampa Scale of Kinesiophobia (TKS) with scores ranging from 17 to 68. Higher scores indicate higher degree of kinesiophobia.

CONTACTS AND LOCATIONS:
Overall Officials: Paula Camargo, PhD, Study Director — Universidade Federal de Sao Carlos
Locations (1):
- Universidade Federal de São Carlos, São Carlos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kamonseki DH, Haik MN, Ribeiro LP, Almeida RF, Camargo PR. Scapular movement training is not superior to standardized exercises in the treatment of individuals with chronic shoulder pain and scapular dyskinesis: randomized controlled trial. Disabil Rehabil. 2023 Sep;45(18):2925-2935. doi: 10.1080/09638288.2022.2114552. Epub 2022 Aug 24. PMID 36000960
- [Derived] Kamonseki DH, Haik MN, Camargo PR. Scapular movement training versus standardized exercises for individuals with chronic shoulder pain: protocol for a randomized controlled trial. Braz J Phys Ther. 2021 Mar-Apr;25(2):221-229. doi: 10.1016/j.bjpt.2020.08.001. Epub 2020 Aug 18. PMID 32855073